CLINICAL TRIAL: NCT03152435
Title: Phase I/II Study of EGFR CART Cells for Patients With Metastatic Colorectal Cancer.
Brief Title: EGFR CART Cells for Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: The Beijing Pregene Science and Technology Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstShenzhen02
Record Dates: First submitted 2017-05-07; First posted 2017-05-15 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-05

CONDITIONS: EGFR-positive Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-tumor response of CART-EGFR (Experimental)
  Interventions: Biological: EGFR CART

INTERVENTIONS:
Biological: EGFR CART — EGFR CART cells will be administered using a split dose on day0 (10%),1(30%), and 2(60%).

SUMMARY:
This is a clinical study to observe the maximum tolerated dose (MTD) and the safety and feasibility of chimeric antigen receptor EGFR (EGFR CART) cells in metastatic patients with colorectal cancer.

DETAILED DESCRIPTION:
This is a study for the patients with colorectal cancer. Maximum tolerated dose climbing test is expected into the group of 9 cases of patients. And Phase II expected into the group of 11 subjects, selected the above safe dose, carrying out a research into the clinical effectiveness. Subjects will be collected their T cells and modify them, the modification is a genetic change, that EGFR:4-1BB:CD28:CD3 modified T cells, in order to tells the T cells to recognize their target tumor cells and potentially kill them, but not other normal cells in the subject's body. The CART cells will then be expanded in vitro and then administered to subjects. The purpose of this study is observe the MTD and to assess the safety and feasibility of CART cells in the patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be 18 years to 70 years;
* 2. Clinical diagnosis of EGFR positive for patients with metastatic colorectal cancer;
* 3. Patients must have a KPS of >80, expected survival > 3 months;
* 4. Patients must have at least one measurable lesions;
* 5. Recently did not use glucocorticoid;
* 6. Patients must have evidence of adequate hepatic and renal function as evidenced by the following laboratory parameters: WBC ≥ 4.0×109/L, Hb ≥90 g/L, PLT ≥100×109/L）; AST ≤2.5ULN，ALT ≤ 2.5ULN; Cr≤ 3ULN; TBIL≤ 3ULN，
* 7. Patients must have a good heart function (LVEF>50%) ;
* 8. Patients must be willing to practice birth control during and for three months following treatment.NOTE:female participants of reproductive potential must have a negative serum pregnancy test, and willing to practice birth control during and for three months following treatment；
* 9. Patients must be willing to sign an informed consent.

Exclusion Criteria:

* 1. Patients with other cancer history;
* 2. Patients allergic to cetuximab;
* 3. Patients with severe bronchitis, bronchial asthma, or severs pneumonia;
* 4. Patients with uncontrolled active infections (bacteria, viruses or fungi infection) ;
* 5. Patients with acute and chronic GVHD (graft versus host disease)
* 6. Patients with severe autoimmune diseases;
* 7. Previously treatment with T cell inhibitors (cyclophosphamide, FK506);
* 8. Patients with active hepatitis B or hepatitis C infection, HIV infection, syphilis serology reaction positive;
* 9. Patients who are participating or participated any other clinical research in the past 1 months;
* 10. Pregnant and/or lactating women will be excluded;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events as assessed by CTCAE v4.0 | 24 weeks

SECONDARY OUTCOMES:
Anti-tumor responses to EGFR CART cells in vivo. | 24 weeks
Determine duration of in vivo survival of EGFR CART . | 1 year
  EGFR CART vector sequences will be determined by Q-PCR

CONTACTS AND LOCATIONS:
Overall Officials: geng tian, Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- The Second People's Hospital of Shenzhen, Shenzhen, Guangdong, China